CLINICAL TRIAL: NCT04355299
Title: Effectiveness of a Short-term Mixed Exercise Program for Treating Sarcopenia in Hospitalized Patients Aged 80 Years and Older
Brief Title: A Short-term Mixed Exercise for Sarcopenic Hospitalized Aged 80+ Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuxiang Liang (Other)
Responsible Party: Sponsor-Investigator, Yuxiang Liang, Physiotherapist, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019#611#
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): a mixed exercise program including aerobic, balance, and resistance exercises that were personally tailored.
  Interventions: Behavioral: balance training; Behavioral: resistance training; Behavioral: aerobic exercise
- control group (Other): usual care
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: balance training — The training to improve balance is to work on the core muscle groups that help to maintain your posture.,and increase muscular strength.
  Arms: Intervention group
Behavioral: resistance training — Resistance training is a form of exercise that improves muscular strength and endurance. During a resistance training workout, you move your limbs against resistance provided by your body weight, gravity, bands, weighted bars or dumbbells.
  Arms: Intervention group
Behavioral: aerobic exercise — Aerobic exercise is any activity that gets your blood pumping and large muscle groups working. It's also known as cardiovascular activity.
  Arms: Intervention group
Behavioral: usual care — received usual care
  Arms: control group

SUMMARY:
Most previous clinical trials that addressed exercise for sarcopenic elderly subjects focused on community-dwelling older adults who were relatively healthy. There is a notable paucity of high-quality research investigating the effects and feasibility of exercise for hospitalized or institutionalized older people, who are generally frailer and more severe in functional impairment than those living in the community. Moreover, most reported exercise programs were of long-term duration, which typically lasted 3 to 6 months with two sessions per week. It remains unclear whether short-term exercise would be effective for treating sarcopenia. Therefore, the investigators aimed to assess the effectiveness of short-term exercise for treating sarcopenia in hospitalized older patients aged 80 years and over.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥80 years;
2. being able to ambulate (assistance was acceptable);
3. being able to communicate and collaborate with the physiotherapist;
4. with sarcopenia defined by the AWGS criteria ;

Exclusion Criteria:

1. terminal illness;
2. uncontrolled heart failure;
3. myocardial infarction within the past three months;
4. uncontrolled respiratory failure;
5. bone fractures within the past three months;
6. acute pulmonary embolism;
7. major surgery within the past three months;
8. uncontrolled arrhythmia;
9. refusal to participate in this study.

Ages: 80 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The change of activities of daily living from the baseline to the end of the 2-week intervention | 2 weeks
  Basic activities of daily living (BADL) assessed by Barthel Index. The total score for Barthel Index ranges from 0 (worst) to 100 (best) points.

SECONDARY OUTCOMES:
The change of gait speed | 2 weeks
  Gait speed was measured using a 4-meter walking test.
The change of handgrip strength | 2 weeks
  Handgrip strength was measured using a digital grip dynamometer
The change of the score of Short Physical Performance Battery | 2 weeks
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. The total score for SPPB ranges from 0 (worst) to 12 (best) points.
The change of the score of Timed Up and Go test | 2 weeks
  The Timed Up and Go test (TUG) is a simple test used to measure basic functional mobility and safety with mobility. The score for the TUG is the time consumption of the whole process. The longer time consuption indicates the more worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiaojiao Jiang, Principal Investigator — West China Hospital; Ming Yang, Study Director — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided